CLINICAL TRIAL: NCT03749746
Title: Heart Health 4 New Moms: A Randomized Controlled Trial of a Lifestyle Intervention and Home Blood Pressure Monitoring Following Preeclampsia in Overweight and Obese Women
Brief Title: Heart Health 4 New Moms: A Randomized Trial in the First Year After Preeclampsia
Acronym: HH4NM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Alisse Hauspurg, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18080007
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Preeclampsia; Gestational Hypertension; Hypertension; Obesity; Overweight and Obesity; Pregnancy Complications; Pregnancy Toxemia; Postpartum Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Hypertension; Obesity; Overweight; Pregnancy Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (Active Comparator): Participants will be counseled on routine postpartum care and will receive additional information on cardiovascular risk following preeclampsia as well as information on support groups and registries as well as online resources for lifestyle modification.
  Interventions: Other: Usual care
- Home Blood Pressure Monitoring (Experimental): In addition to usual care outlined above, each participant will receive a Bluetooth-enabled blood pressure cuff along with a checklist of proper technique and instructions on use. Women will be prompted to measure their BP across the first week of each month during the intervention. Based on guidelines, participants will take their blood pressure in the morning and evening, each time taking two readings separated by one minute.
  Interventions: Behavioral: Home Blood Pressure Monitoring
- Heart Health 4 New Moms (Experimental): Participants randomized to this group will receive instruction on the use of Heart Health 4 New Moms internet-based lifestyle intervention and home blood pressure monitoring. The internet-based intervention is comprised of four key components: an online curriculum with modules on healthy eating and physical activity, a self-monitoring and tracking program, a registered dietitian will act as a lifestyle coach for participants and a customized online toolbox.
  Interventions: Behavioral: Home Blood Pressure Monitoring; Behavioral: Heart Health 4 New Moms

INTERVENTIONS:
Behavioral: Home Blood Pressure Monitoring — Each participant will receive 1:1 training by the project staff in all aspects of home blood pressure monitoring (HBPM). Throughout the study, they will be asked to monitor home blood pressures for the first week of each month with Bluetooth-enabled blood pressure cuffs.
  Arms: Heart Health 4 New Moms; Home Blood Pressure Monitoring
Behavioral: Heart Health 4 New Moms — The intervention is comprised of four key components: (1) The online curriculum consists of 12 modules on healthy eating and physical activity adapted from the Diabetes Prevention Program and specifically targeting postpartum women. (2) Self-monitoring and tracking program, in which participants will be provided with a Bluetooth-enabled blood pressure cuff and digital scale and will be provided real-time feedback on their blood pressure and weight trends. (3) A registered dietitian will act as a lifestyle coach for participants with regular review of progress and provision of coaching notes, support and suggestions. (4) Finally participants will have access to a customized online toolbox, including dietary tracking sheets and recipes from the American Heart Association (AHA).
  Arms: Heart Health 4 New Moms
Other: Usual care — Participants will be counseled on routine postpartum care and will receive additional information on cardiovascular risk following preeclampsia as well as information on support groups and registries as well as online resources for lifestyle modification.
  Arms: Usual care

SUMMARY:
Preeclampsia causes devastating maternal and neonatal morbidity and mortality with a high recurrence risk and a rapid, occult progression to cardiovascular disease after delivery. There is a critical need for effective interventions to reduce these risks. This is a pilot randomized controlled trial of a novel postpartum lifestyle intervention compared to women who take home blood pressure measurements and women with usual care who are overweight and obese in the first year after preeclampsia. The investigators hypothesize that the intervention will lead to improved weight loss and blood pressure in the first year postpartum, which has broad implications for future pregnancy and long-term cardiovascular health.

DETAILED DESCRIPTION:
The overall objective of this study is to conduct a pilot trial of an internet-based lifestyle intervention and home blood pressure monitoring in the year after delivery among overweight and obese women with preeclampsia to evaluate feasibility, acceptability and to assess the effect of the intervention. The investigators hypothesize that compared to usual care, an internet-based lifestyle intervention implemented in the immediate postpartum period in overweight and obese women with preeclampsia improves weight loss at one year postpartum. 150 overweight or obese women with preeclampsia will be randomized into internet-based lifestyle intervention plus home blood pressure monitoring, home blood pressure monitoring alone, or usual care groups in the postpartum period. The investigators will assess feasibility by the proportions of women who are eligible, enroll, and remain in the study at one year. The effect of home blood pressure monitoring on blood pressure and progression to sustained hypertension will also be explored. A successful outcome of this study would have a direct impact to improve cardiovascular health and future pregnancy health in women who have had preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* pre-pregnancy body mass index ≥25 kg/m2
* diagnosed with preeclampsia or gestational hypertension
* access to internet

Exclusion Criteria:

* multiple gestation
* medical co-morbidities: chronic kidney disease, active liver disease (acute hepatitis, chronic active hepatitis), active cardiac disease, pre-pregnancy diabetes mellitus, chronic hypertension diagnosed prior to pregnancy
* pregnancy prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-01-26 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Weight loss | 4-8 weeks postpartum to 8-12 months postpartum
  weight change between two study visits

SECONDARY OUTCOMES:
Systolic blood pressure | 8-12 months postpartum
  Systolic blood pressure at study visit 2
Diastolic blood pressure | 8-12 months postpartum
  Diastolic blood pressure at study visit 2
Hypertension | 8-12 months postpartum
  Proportion of women with hypertension by AHA guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Alisse Hauspurg, MD, Principal Investigator — Magee-Womens Hospital of University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hauspurg A, Bryan S, Jeyabalan A, Davis EM, Hart R, Shirriel J, Muldoon MF, Catov JM. Blood Pressure Trajectories Through the First Year Postpartum in Overweight or Obese Individuals Following a Hypertensive Disorder of Pregnancy. Hypertension. 2024 Feb;81(2):302-310. doi: 10.1161/HYPERTENSIONAHA.123.22231. Epub 2023 Dec 11. PMID 38073563